CLINICAL TRIAL: NCT07145411
Title: HPC Offered for PRESERVE Expansion
Acronym: HOPE
Status: Recruiting | Type: Observational
Sponsor: Ossium Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HOPE Program; HOPE (Other: Ossium Health)
Record Dates: First submitted 2025-07-10; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Bone Marrow Transplant (BMT)
Keywords: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Lymphomas; Chronic lymphoblastic Leukemia; Chronic Myeloid Leukemia; myelodysplastic syndrome; stem cell transplant; severe aplastic anemia; Sickle cell anemia; Thalessemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Anemia, Aplastic; Anemia, Sickle Cell | interventions — Bone Marrow Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ossium HPC, Marrow: Ossium HPC, Marrow will be provide for infusion on the day of transplant
  Interventions: Other: Bone Marrow Transplant with Ossium's HPC, Marrow (bone marrow recovered from deceased organ and tissue donors)

INTERVENTIONS:
Other: Bone Marrow Transplant with Ossium's HPC, Marrow (bone marrow recovered from deceased organ and tissue donors) — The HOPE Program does not include any investigational drugs. The medicines and procedures in this program are standard of care for a transplant. Bone marrow cells from a deceased organ and tissue donor for use in your transplant is the only product offered to you by Ossium Health.

SUMMARY:
Ossium recognizes that not all patients who could benefit from Ossium's HPC, Marrow can access the PRESERVE trial for logistical or eligibility reasons. The HOPE program is expanded access program to serve these patients by providing our bone marrow product

ELIGIBILITY:
Inclusion Criteria:

Patients aged 12-80 may be eligible* to receive bone marrow for transplantation through the Ossium HOPE Program if:

Their treating physician determined they are eligible for allogeneic bone marrow transplant Their treating physician determined that the potential benefit outweighs the potential risks

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing allogenic bone marrow transplant
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Neutrophil engraftment | 28 days
  1. To determine cumulative incidences of neutrophil engraftment (ANC ≥500/µL for 3 consecutive values)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Henry Ford Health, Detroit, Michigan
  - The Ohio State University Medical Center, Columbus, Ohio
  - Tristar Centennial Medical Center, Nashville, Tennessee